CLINICAL TRIAL: NCT03477773
Title: Development of an Exergame to Deliver a Sustained Dose of High-Intensity Training: Formative Pilot Randomized Trial
Brief Title: Development of an Exergame to Deliver a Sustained Dose of High-Intensity Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Teesside University (Other); Northumbria University (Other); Newcastle University (Other)
Responsible Party: Principal Investigator, Tom McBain, Principal Investigator, Sheffield Hallam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SheffieldHU
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Metabolic Syndrome
Keywords: high-intensity interval training; video games; heart rate; boxing; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Pilot, exploratory, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Perform three session of high-intensity, interval training sessions per week over the 6-week intervention
  Interventions: Other: High-intensity exergaming
- Control (No Intervention): Continue with their normal habitual lifestyle over the 6-week intervention

INTERVENTIONS:
Other: High-intensity exergaming — Perform high-intensity exercise whilst playing a developed exergame. A full warm-up performed prior to the session was performed (~70% HRmax). Periods of exercise were performed at an intensity >85% HRmax for periods of 10, 20 and 30s, interspersed with periods of rest, for a total of 2-3 minutes per session. Heart rate was monitored throughout the intervention.
  Arms: Intervention

SUMMARY:
Males from areas of social deprivation within the town of Middlesbrough (UK) were targetted and recruited on to a high-intensity, exergaming intervention over a 6-week period. Eligible participants were randomly allocated to an intervention group (weekly exergaming) or control group (normal habitual lifestyle). All participants completed baseline (week 0) and follow-up (week 7) measures of metabolic health. Participants in the intervention group were invited to three sessions a week of high-intensity exergaming performed against their peers on a developed boxing game.

DETAILED DESCRIPTION:
A 6-week exploratory controlled trial designed to assess the fidelity of the game in terms of delivering the intended training stimulus and to examine the effect of the intervention on selected health outcomes was conducted. As appropriate for an exploratory trial, the investigators did not conduct formal sample size estimation a priori, rather the CIs would be used to inform future trials. A targeted recruitment approach at locations predominantly attended by men may facilitate uptake of participants was used. Therefore, to maximize recruitment within the intended population, relevant gatekeepers were approached at institutions positioned within regions of social deprivation. Thus, two settings used for recruitment and the trials were a social club and mosque, both situated within deprived regions of Middlesbrough, United Kingdom (TS1 and TS4). A total of 24 males were recruited into the trial (Figure 4) using relevant gatekeepers at institutions positioned within regions of social deprivation. Two recruitment drives (October 2014 and February 2015) took place, and these involved live demonstrations of the technology followed by word-of-mouth and snowballing approaches. The exergaming system was important in this recruitment process because it provided something tangible and interesting to engage potential participants.

A third-party minimization process using baseline measures of age, waist circumference, and predicted maximum oxygen consumption (VO2 max) was used to remove bias in group allocation. The control group was instructed to maintain their current physical activity levels and inform the researchers should any changes arise during the intervention period. Overall retention to the intervention that encompassed baseline and follow-up measures was 87.5% (21/24).

To explore perceptions of the exergame and the HIT regime, semistructured interviews were conducted with 5 intervention participants following the 6-week training period, which were analyzed semantically. The study was approved by the ethics committee of Teesside University, United Kingdom, and written informed consent was obtained from all participants.

Evidence recommends a minimum duration of 12 weeks for a HIT protocol to promote favorable changes in blood pressure and anthropometric measurements of obesity [35]. However, a 6-week intervention was selected, as a minimum of 13 sessions (0.16 work/rest ratio) is sufficient to elicit moderate improvements in VO2 max in sedentary individuals. Additionally, there is still ambiguity regarding the optimal work-to-rest ratio when designing HIT interventions, particularly in populations with varied age, baseline fitness, and training experience. Therefore, longer duration HIT models (1-4 min) were deemed unsuitable for the target population. Furthermore, minigames (such as the current exergame) have short life spans, where adherence to a longer intervention (eg, 12 weeks) may diminish over time and influence health outcomes. This was evident from a 12-week pilot study (unpublished data) using an exergame in the same population that saw attendance drop from 53% during week 2 to 16% during week 12.

Participants allocated to the intervention group were invited to attend three sessions of exergaming per week. At the beginning of the exergaming session, participants were required to complete a 6-min structured warm-up consisting of a series of exercises on a 210 mm step until both participants reached >70% HRmax. Session workloads with volumetric progression were set automatically once the user's identifying information was entered. The session workloads were 120-s, 150-s, and 180-s of work during weeks 1 and 2, weeks 3 and 4, and weeks 5 and 6, respectively.

To avoid staleness, the repetition lengths (10, 20, or 30-s) were randomly selected at the beginning of each round. The investigators set the work-to-rest ratio at 1:4, and thus, the respective repetitions were followed by 40, 80, or 120-s of active recovery. Participants were instructed to perform the repetitions at an intensity ≥85% HRmax. Each exergaming session took approximately 30 to 40 min to complete, including equipment set-up, warm-up with additional enjoyment, and task immersion questionnaires upon completion of the HIT bouts (not reported here). Heart rate responses were taken within repetitions and therefore, did not include any of the recovery period. This, therefore, avoided an overestimation of physiological load, which can occur when heart rate continues to rise after exercise cessation.

ELIGIBILITY:
Inclusion Criteria:

* 'apparently healthy' according the ACSM guidelines

Exclusion Criteria:

* known presence of cardiovascular disease
* musculoskeletal injury

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males only
Enrollment: 24 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Six-weeks
  Predicted VO2max was obtained by performing a submaximal 8-min ramped step test. Heart rate response (Polar T34; PolarElectro OY, Kempele, Finland) and simultaneous breath-by-breath expired gas were collected using a portable indirect calorimeter (Cosmed K4 b2; Rome, Italy), calibrated per the manufacturer's guidelines. Individual HRmax was estimated and plotted against VO2 data for the determination of predicted VO2max (reported in ml.kg.min-1).
Blood pressure | Six-weeks
  Blood pressure was collected on the left arm positioned at heart height with the subjects in a seated position by an automatic upper arm blood pressure monitor (Omron MX13). Measures were made at least three times at 3-min intervals, where an average of the two lowest measures was used for analysis (reported in mm/Hg).
Waist circumference | Six-weeks
  Waist circumference was measured using the World Health Organization guidelines (reported in cm).
Body Mass | Six-weeks
  Body mass was measured using a portable set of electronic scales (Seca, Birmingham, UK) and reported the neasrest 0.1kg.

SECONDARY OUTCOMES:
Within-participant heart rate | Six-weeks
  To observe the within-participant heart rate responses to the 10, 20 and 30s high-intensity repetitions across the intervention (reported as percentage of individual heart rate maximum (%).
Between-participant heart rate | Six-weeks
  To observe the between-participant heart rate responses to the 10, 20 and 30s high-intensity repetitions across the intervention (reported as percentage of individual heart rate maximum (%).

OTHER OUTCOMES:
Perceptions of the high-intensity exergame | Six-weeks
  Semistructured interviews were conducted with intervention participants following the 6-week training period to explore the feasability of the intervention and developed exergame

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD from the current study.

REFERENCES:
- [Derived] McBain T, Weston M, Crawshaw P, Haighton C, Spears I. Development of an Exergame to Deliver a Sustained Dose of High-Intensity Training: Formative Pilot Randomized Trial. JMIR Serious Games. 2018 Mar 27;6(1):e4. doi: 10.2196/games.7758. PMID 29588271

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03477773/Prot_SAP_ICF_000.pdf